CLINICAL TRIAL: NCT00006167
Title: Nutrition Intervention in AIDS Wasting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: NIAW (completed); DK51011
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: HIV Wasting Syndrome
Keywords: oxandrolone; AIDS wasting; strength training; progressive resistance training; exercise; dietary intervention
MeSH Terms: conditions — HIV Wasting Syndrome; Motor Activity | interventions — Oxandrolone

INTERVENTIONS:
Drug: oxandrolone
Behavioral: Progressive Resistance Training

SUMMARY:
There are no guidelines for appropriate nutritional management of weight loss or wasting in HIV infection. Some treatments may increase weight, but without improving muscle mass or quality of life. In this clinical trial AIDS patients with wasting are randomized to one of three nutritional strategies and studied over a 12-week period: 1) optimal oral nutrition with counseling and protein and calorie supplementation, and a placebo pill; 2) optimal oral nutrition with the oral androgen, oxandrolone at 20 mg daily; and 3) optimal oral nutrition with progressive resistance training (PRT). In all participants, dietary intervention is maximized by weekly personalized counseling to address individual issues and concerns. Two primary outcomes are assessed: thigh muscle mass and quality of life. Our findings can be used to develop guidelines for standards of nutritional care among AIDS patient with the wasting syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Loss of 10% of usual body weight, OR loss of 5% of usual body weight within the previous 6 months, OR BMI20kg/m2. If the candidate is taking a protease inhibitor, he/she must have not regained weight since initiating the medication over a period of at least 4 weeks prior to screening.
* Documented HIV-positive
* Able to eat
* English-speaking
* Compliance with medical regimens
* For heterosexually active women: willingness to use an effective means of birth control
* Patient and physician not planning to start new treatments for HIV infection or weight loss during the 12 weeks of study.

Exclusion Criteria:

* Vomiting 1 time/day or diarrhea 4 times/day on average in the previous week
* Fever 101 F within the previous week
* Receiving induction treatment for one of the following (new diagnosis or recurrence within 4 weeks):

Pneumocystis carinii pneumonia Cryptococcal meningitis Cytomegalovirus retinitis or pneumonitis Toxoplasmosis Mycobacterium avium complex Visceral Kaposi's Sarcoma Lymphoma Pulmonary tuberculosis

* Received corticosteroids, estrogens, progesterones, androgens, oral anticoagulants, or growth hormone within the previous three months
* History of life-threatening reaction to oxandrolone or testosterone
* Currently pregnant
* History of congestive heart failure, myocardial infarction, angina/coronary artery disease, uncontrolled hypertension, cerebrovascular accident, hepatic failure, bleeding disorder, diabetes, nephrotic syndrome, cancer of the breast or prostate, or hypercalcemia
* Milk product allergy
* Current use of injected drugs
* Participation in an exercise program or strength training within the previous 4 weeks
* Any medical condition which renders the participant physically incapable of performing strength exercises
* Serum total testosterone level at least 300ng/ml, unless patient and primary physician prepared to begin testosterone injections concurrent with study enrollment (men only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-01; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Gorbach, MD, Principal Investigator — Tufts University; Abby Shevitz, MD, Study Director — Tufts University
Locations (1):
- Tufts University School of Medicine, Boston, Massachusetts, United States